CLINICAL TRIAL: NCT07164950
Title: A Multicenter, Prospective, Phase II Clinical Trial Investigating the Use of Compression Stockings to Prevent Peripheral Neuropathy Induced by Antibody-Drug Conjugates (ADCs) in Patients With Urothelial Carcinoma
Brief Title: Compression Stockings to Prevent Peripheral Neuropathy Caused by Antibody-Drug Conjugates in Urothelial Carcinoma Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sheng Zhang (Other)
Responsible Party: Sponsor-Investigator, Sheng Zhang, Prof., Fudan University
Organization: Fudan University (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: CIPN-ADC-002
Record Dates: First submitted 2025-08-10; First posted 2025-09-10 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Urothelial Carcinoma; Advanced Solid Tumors; Chemotherapy-Induced Peripheral Neuropathy; Antibody-drug Conjugates
Keywords: Antibody-Drug Conjugates; Peripheral Neuropathy Prevention; Compression Stockings; Advanced Cancer; Quality of Life; Mechanical Compression Therapy
MeSH Terms: conditions — Carcinoma, Transitional Cell

STUDY DESIGN:
Intervention Model Description: Self-controlled, within-subject comparison: left foot receives compression stocking, right foot serves as control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Compression Stocking Arm (Experimental): Each participant will wear a medical-grade compression stocking (Class II, 20-30 mmHg) on the assigned foot throughout the entire treatment period with antibody-drug conjugates (ADCs). Stockings are worn daily except during bathing.
  Interventions: Device: Medical-grade compression stocking
- Control Arm (No Stocking) (No Intervention): The contralateral foot will not receive any compression stocking and will be observed under the same ADC treatment conditions. Each participant serves as their own control.

INTERVENTIONS:
Device: Medical-grade compression stocking — A knee-high compression stocking providing 20-30 mmHg pressure will be applied to the assigned foot during the ADC treatment period to prevent chemotherapy-induced peripheral neuropathy (CIPN). Stockings will be worn daily, except during bathing.
  Arms: Compression Stocking Arm

SUMMARY:
This multicenter, prospective phase II clinical trial aims to evaluate the efficacy and safety of medical compression stockings in preventing peripheral neuropathy induced by antibody-drug conjugates (ADCs) containing monomethyl auristatin E (MMAE) in patients with advanced cancers, including urothelial carcinoma. Eligible participants will have no baseline ≥ grade 1 neuropathy and will be scheduled to receive MMAE-containing ADC therapy. A total of 58 patients will be enrolled and followed for 24 months. In this self-controlled design, the left foot will be fitted with a medical compression stocking while the right foot remains uncovered, starting 15 minutes before infusion and continuing until 15 minutes after infusion (total duration: 120 minutes). Peripheral neuropathy will be assessed before treatment, after cycle 3, within 1 week after treatment completion, and 1 month after completion, using CTCAE v5.0 and patient-reported questionnaires (QLQ-C30 and FACT-GOG-NTx). Toe temperature will be measured to assess local microcirculation changes. The study will also monitor compression-related adverse events. The results will provide evidence for preventive strategies to reduce ADC-induced peripheral neuropathy and improve patients' quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years Histologically or cytologically confirmed advanced malignancy (including but not limited to urothelial carcinoma) eligible for MMAE-containing ADC therapy (e.g., EV, DV, BV)
* ECOG performance status 0-2
* No baseline peripheral neuropathy ≥ Grade 1 (CTCAE v5.0)
* Stable tumor status without other neurotoxic drugs in the past 2 months
* Adequate organ function (blood counts, liver and kidney function) per protocol
* Expected survival ≥ 3 months
* Ability and willingness to comply with study procedures and provide written informed consent

Exclusion Criteria:

* Poor compliance or inability to follow protocol
* Pre-existing peripheral neuropathy ≥ Grade 1 from prior platinum/taxane treatment
* Severe diabetes or peripheral vascular disease
* Neurological disorders causing nerve compression (e.g., carpal tunnel syndrome, radiculopathy)
* Severe psychiatric conditions (depression, bipolar disorder, substance abuse)
* Active uncontrolled infections requiring systemic antibiotics/antifungals/antivirals (≥ CTCAE Grade 2)
* Active hepatitis or significant liver dysfunction not meeting inclusion criteria
* Renal failure requiring dialysis
* Immunodeficiency or history of organ transplantation
* Severe nausea, headache, fatigue, or other debilitating symptoms
* Active tuberculosis or uncontrolled pleural/pericardial effusion/ascites
* Hypersensitivity to monoclonal antibodies or study device components
* Participation in other clinical trials within 4 weeks
* Known bleeding or coagulation disorders or receiving thrombolytic therapy
* Any other condition judged by the investigator to preclude safe participation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2025-08-30 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Grade ≥1 Peripheral Neuropathy (CTCAE v5.0) | Baseline (within 7 days before treatment start); At the end of Cycle 3 (each cycle = 28 days, within 7 days); At treatment completion (within 7 days of last ADC dose); 1 month (±7 days) after treatment completion.
  The proportion of patients who develop Grade ≥1 peripheral neuropathy, as assessed by CTCAE version 5.0.

SECONDARY OUTCOMES:
Change in Quality of Life Scores (EORTC QLQ-C30) | Baseline; At the end of Cycle 3 (each cycle = 28 days); At treatment completion (within 7 days of last ADC dose); 1 month (±7 days) after treatment completion.
  Change in patient-reported quality of life assessed using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30). Scores range from 0 to 100; higher scores indicate better quality of life.
Peripheral Neuropathy Severity (FACT-GOG-NTx Scale) | Baseline; At the end of Cycle 3 (each cycle = 28 days); At treatment completion (within 7 days of last ADC dose); 1 month (±7 days) after treatment completion.
  Severity of chemotherapy-induced neuropathy symptoms assessed by the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity (FACT-GOG-NTx) subscale. Scores range from 0 to 44; higher scores indicate more severe neuropathy.
Left vs. Right Lower Limb Neuropathy Comparison (FACT-GOG-NTx Scale) | Baseline; At the end of Cycle 3 (each cycle = 28 days); At treatment completion (within 7 days of last ADC dose); 1 month (±7 days) after treatment completion
  Assessment of lower limb neuropathy symptoms, focusing on sensory and motor impairment, using a 4-item subscale from the FACT-GOG-NTx questionnaire. Each item is scored from 0 to 4, with total scores ranging from 0 to 16; higher scores indicate more severe neuropathy.
Incidence of Grade ≥2 Peripheral Neuropathy (CTCAE v5.0) | Measured at baseline, after the 3rd treatment cycle, at treatment completion, and 1 month after treatment completion.
  Proportion of patients developing Grade 2 or higher peripheral neuropathy as per CTCAE 5.0 criteria.
Toe Temperature Changes (Infrared Thermography) | Baseline (within 7 days before treatment start); At the end of Cycle 3 (each cycle = 28 days, within 7 days).
  Change in toe temperature measured using infrared thermography, as an indicator of local microcirculation changes.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China